CLINICAL TRIAL: NCT04294550
Title: A Multicenter, Observational Prospective Study on Quality of Life (QOL) in Advanced Cancer Patients With Opioid-induced Constipation (OIC) Treated at Home With Naloxegol According to the Clinical Practice
Brief Title: Study on Quality of Life in Advanced Cancer Patients With Opioid-induced Constipation Treated With Naloxegol
Status: Completed | Type: Observational
Sponsor: Fondazione ANT Italia ONLUS (Other)
Responsible Party: Sponsor
Other Study IDs: 293/2018/OSS/AUSLBO
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Opioid Use; Constipation Drug Induced; Cancer
Keywords: Opioid induced constipation; Cancer patients; Palliative care; Quality of life; PAC-QoL; Naloxegol
MeSH Terms: conditions — Neoplasms; Opioid-Induced Constipation | interventions — naloxegol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Naloxegol — 28 days of therapy with 25 mg/day of Naloxegol on cancer patients using opioids and suffering for opioids induced constipation not relieved by first-line laxatives.

SUMMARY:
Opioid-Induced Constipation (OIC) is often associated with a compromised quality of life of patients in palliative care (PC) setting. Among the Peripherally-Acting Mu-Opioid Receptor Antagonists, Naloxegol is the most effective to treat OIC and to improve OIC-related aspects of quality of life in patients with non-cancer pain.

This observational study aims to assess the impact of a 4-weeks Naloxegol therapy on the quality of life in advanced cancer patients with OIC assisted by a home PC program.

The study is enrolling cancer patients with OIC (defined according to Rome IV criteria) not relieved by first-line laxatives, starting the therapy with 25 mg/day of Naloxegol. The main parameters evaluated at the beginning of the therapy (T0) and after 28 days (T28) are: Patient Assessment of Constipation Quality-of-Life (PAC-QoL, 4 subscales: physical discomfort, psychosocial discomfort, worries and concerns, satisfaction), evaluation of objective (number of weekly evacuations) and subjective constipation (Bowel Function Index, BFI, normal score<30), pain assessment by NRS.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients with advanced disease;
* age higher than 18 years;
* mentally competent;
* naloxegol therapy for no more than 1 week according to clinical practice;
* sign of a written informed consent.

Exclusion Criteria:

* patient with pain not controlled by opioids;
* therapy with other PAMORAs;
* intestinal obstruction;
* risk of intestinal perforation.
* severe renal failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients with constipation induced by opioids who do not respond to the usual laxatives, under naloxegol therapy (25mg/day) assisted at home by the palliative care program of Fondazione ANT Italia ONLUS.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Patient Assessment of Constipation Quality-of-Life (PAC-QoL) score | 4 weeks
  Change of quality of life evaluated by Patient Assessment of Constipation Quality-of-Life (PAC-QoL) at T0 and T28. Each item of the 28-item questionnaire was scored on a 5-point Likert-type scale from 0 to 4, with (0 = none/not at all, 1 = a little bit/a little bit of the time, 2 = moderately/some of the time, 3 = quite a bit/most of the time, 4 = extremely/all the time). Scores were reported overall and for each of the four subscales (physical discomfort, psychosocial discomfort, worries and concerns, and satisfaction). An improvement (reduction) of ≥1 point in PAC-QOL score was considered clinically significant based on previous validation studies.

SECONDARY OUTCOMES:
Objective constipation | 4 weeks
  Change of objective constipation evaluated by number of weekly evacuations.
Subjective constipation | 4 weeks
  Change of subjective constipation evaluated by Bowel Function Index (BFI). The BFI is a physician-administered, patient-assessment scale made up of three items: (1) ease of defecation, (2) feeling of incomplete bowel evacuation, and (3) personal judgement of constipation during the last 7 days. The physician asks the patient to rate his or her impression of each of the three items during the previous week on a scale from 0 to 100, with 0 signifying 'not at all' and 100 signifying 'very strong'. The score is then calculated as the average of the three components of the scale with each component being weighted equally. The BFI total score remains on a scale of 0 to 100 with higher scores indicating greater constipation.
Pain (Numeric Rating Scale) | 4 weeks
  Change of pain assessed by Numeric Rating Scale (NRS). The NRS is a 11-points numeric scale through participants were asked to rate their average pain intensity by selecting a single number from 0 to 10. Higher scores indicate a more severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Ruggeri, MD, Principal Investigator — Fondazione ANT Italia ONLUS
Locations (1):
- Fondazione ANT Italia ONLUS, Bologna, BO, Italy

REFERENCES:
- [Result] Ostan R, Gambino G, Malavasi I, Ronga G, Solipaca M, Spunghi M, Varani S, Pannuti R, Ruggeri E. Can Naloxegol Therapy Improve Quality of Life in Patients with Advanced Cancer? Cancers (Basel). 2021 Nov 16;13(22):5736. doi: 10.3390/cancers13225736. PMID 34830889